CLINICAL TRIAL: NCT06137131
Title: Voice Therapy With a Semi-occluded Vocal Tract: From Current Challenges to Next Level Efficacy Studies
Brief Title: Voice Therapy With a Semi-occluded Vocal Tract
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Research Foundation Flanders (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 249721N
Record Dates: First submitted 2023-10-20; First posted 2023-11-18 (Actual); Results first posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-08

CONDITIONS: Voice Disorders
Keywords: voice; semi-occluded vocal tract; larynx; randomized controlled trial; efficacy study
MeSH Terms: conditions — Voice Disorders; Laryngeal Diseases | interventions — Air; Water; Phonation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- straw phonation in air (Experimental): Participants will be asked to phonate an /u/ vowel through a stirring straw in air with slightly pursed lips and a soft voice onset.
  Interventions: Behavioral: Straw phonation in air
- straw phonation in 2 cm water (Experimental): Participants will be asked to phonate an /u/ vowel through a stirring straw, placed 2 cm below the water surface, with slightly pursed lips and a soft voice onset.
  Interventions: Behavioral: straw phonation in water
- straw phonation in 5 cm water (Experimental): Participants will be asked to phonate an /u/ vowel through a stirring straw, placed 5 cm below the water surface, with slightly pursed lips and a soft voice onset.
  Interventions: Behavioral: straw phonation in water
- /u/ control condition (Active Comparator): Participants will be asked to phonate an /u/ vowel with slightly pursed lips and a soft voice onset but without a straw.
  Interventions: Behavioral: /u/ phonation

INTERVENTIONS:
Behavioral: Straw phonation in air — Phonation (/u/ vowel) through a stirring straw (3 mm diameter, 20cm length) in air
  Other Names: steady SOVT exercise
  Arms: straw phonation in air
Behavioral: straw phonation in water — Phonation (/u/ vowel) through a stirring straw (3 mm diameter, 20cm length) in 2 cm or 5 cm water
  Other Names: water-resistance therapy, fluctuating SOVT exercise
  Arms: straw phonation in 2 cm water; straw phonation in 5 cm water
Behavioral: /u/ phonation — /u/ phonation without a straw, control condition
  Other Names: articulatory/steady SOVT exercise
  Arms: /u/ control condition

SUMMARY:
1. The first objective of this research is to investigate the immediate effects of three semi-occluded vocal tract (SOVT) exercises (straw phonation in air, straw phonation in 2cm water, and straw phonation in 5cm water) on (supra)glottic activity of vocally healthy participants and patients with voice disorders (dysphonia) visualized with laryngovideostroboscopy.

   Participants will receive a flexible laryngovideostroboscopy, both during normal phonation and during the specific SOVT exercise. These videos will be randomly and blindly evaluated by two experts using the Voice-Vibratory Assessment with Laryngeal Imaging (VALI) rating form (Poburka et al., 2017).

   Researchers will compare the effects of these SOVT exercises on the (supra)glottic activity with the effects found in a control group producing /u/ phonation, using a randomized controlled trial.
2. The second objective of this research is to investigate the short- and long-term effects of the three SOVT therapy approaches on the (supra)glottic activity, voice quality and self-report of patients with voice disorders (dysphonia).

Participants will receive a short-term intensive therapy with the specific SOVT exercise across four weeks.

Immediately after the therapy program and at 1 and 3 months follow-up, the voice of the participants will be re-evaluated.

ELIGIBILITY:
Patients:

Inclusion criteria are aged between 17 and 50 years, and diagnosed with dysphonia by an otorhinolaryngologist and SLP experienced in voice diagnostics. Exclusion criteria are previous or current participation in voice therapy, previous phonosurgical interventions, pregnancy, smoking, nasal or ear diseases, and neurological disorders.

Vocally healthy participants:

Inclusion criteria are aged between 17 and 50 years. Exclusion criteria are dagnosed with dysphonia, previous or current participation in voice therapy, previous phonosurgical interventions, pregnancy, smoking, nasal or ear diseases, and neurological disorders.

Ages: 17 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 58 (Actual)
Dates: Start 2021-10-07 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2023-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristiane Van Lierde, PhD, Principal Investigator — University Ghent
Locations (1):
- Department of Rehabilitation Sciences, Ghent University (Hospital), Ghent, East-Flanders, Belgium

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Straw Phonation in Air | Straw Phonation in 2 cm Water | Straw Phonation in 5 cm Water | /u/ Control Condition
Started | 15 | 15 | 14 | 14
Completed | 14 | 13 | 13 | 12
Not Completed | 1 | 2 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Straw Phonation in Air | Straw Phonation in 2 cm Water | Straw Phonation in 5 cm Water | /u/ Control Condition | Total
Number analyzed (Participants) | 15 | 15 | 14 | 14 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 14 | 14 | 58
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 18.7 [17 to 20] | 18.7 [17 to 20] | 18.7 [17 to 20] | 18.7 [17 to 20] | 18.7 [17 to 20]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 14 | 14 | 58
  Male | 0 | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 15 | 15 | 14 | 14 | 58
smoking [Count of Participants; unit: Participants] | 1 | 0 | 0 | 0 | 1
organic vocal fold pathology [Count of Participants; unit: Participants] | 0 | 1 | 1 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: (Supra)Glottic Activity: Amplitude of Vibration
Description: Laryngeal function determined with the Voice-Vibratory Assessment with Laryngeal Imaging (VALI) rating form (Poburka et al., 2017).
  Amplitude of vibration: magnitude of lateral movement of the vocal folds. This is a visual-perceptual evaluation based on the video samples of the strobovideolaryngoscopy. Raters score the magnitude of lateral movement of the vocal folds based on the graphic of the VALI form ranging from 0 to 10, this number is then multiplied by 10 to obtain a percentage. Lower percentages mean a smaller amplitude of vibration, higher percentages mean a larger amplitude of vibration.
Time Frame: baseline (before the intervention)
Measure: Mean (Inter-Quartile Range); unit: percentage
Arm/Group | Straw Phonation in Air | Straw Phonation in 2 cm Water | Straw Phonation in 5 cm Water | /u/ Control Condition
Number analyzed (Participants) | 14 | 13 | 13 | 12
percentage
  SOVT phonation | 37.7 [33.6 to 41.7] | 32.5 [28.0 to 37.0] | 28.8 [24.5 to 33.2] | 37.1 [32.6 to 41.6]
  habitual phonation | 36.7 [32.6 to 40.7] | 39.6 [35.1 to 44.1] | 40.0 [35.6 to 44.4] | 34.6 [30.1 to 39.1]

2. Primary Outcome: Supraglottic Activity: Anteroposterior Compression
Description: Laryngeal function determined with the VALI form (Poburka et al, 2017).
  Anteroposterior supraglottic compression: constriction of the supraglottic structures in the anteroposterior dimension. This is a visual-perceptual evaluation based on the video samples of the strobovideolaryngoscopy. Raters score the supraglottic compression based on the graphic of the VALI form on a scale ranging from 0 to 5 (with the aid of concentric circles). The higher the number, the more supraglottic compression. More supraglottic compression is often seen as a negative outcome, however it might be a beneficial effect seen in SOVT phonation studied here.
Time Frame: baseline (before the intervention)
Measure: Mean (Inter-Quartile Range); unit: units on a scale
Arm/Group | Straw Phonation in Air | Straw Phonation in 2 cm Water | Straw Phonation in 5 cm Water | /u/ Control Condition
Number analyzed (Participants) | 14 | 13 | 13 | 12
units on a scale
  SOVT phonation | 2.6 [1.9 to 3.3] | 2.3 [1.4 to 3.1] | 2.9 [2.1 to 3.7] | 1.3 [0.4 to 2.1]
  habitual phonation | 1.2 [0.5 to 1.9] | 1.0 [0.2 to 1.8] | 1.4 [0.7 to 2.2] | 1.4 [0.7 to 2.3]

3. Secondary Outcome: Voice Quality Index 1: Dysphonia Severity Index (DSI)
Description: DSI: A higher index indicates a better voice quality. The index ranges from -5 to +5 for severely dysphonic to normal voices. A more negative index indicates a worse voice quality. Values > +5 are possible in subjects with excellent vocal capacities. A DSI = +1.6 is the threshold separating normophonic from dysphonic persons.
Time Frame: baseline (before the intervention), 1 month (immediately after the intervention), 1 month follow-up, 3 months follow-up
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Straw Phonation in Air | Straw Phonation in 2 cm Water | Straw Phonation in 5 cm Water | /u/ Control Condition
Number analyzed (Participants) | 8 | 8 | 8 | 8
score on a scale
  Baseline | 1.0 [-0.3 to 2.2] | 1.3 [0.0 to 2.5] | 0.7 [-2.5 to 2.0] | 1.0 [-0.3 to 2.2]
  1 month (immediately after the intervention) | 1.7 [0.4 to 3.0] | 1.2 [-0.3 to 2.4] | 0.9 [-0.3 to 2.2] | 0.9 [-0.4 to 2.2]
  1 month follow-up | 2.4 [1.1 to 3.6] | 3.0 [1.7 to 4.4] | 2.3 [1.0 to 3.5] | 1.3 [0.1 to 2.6]
  3 months follow-up | 2.3 [1.1 to 3.6] | 2.5 [1.2 to 3.9] | 1.9 [0.7 to 3.2] | 1.5 [0.1 to 2.9]

4. Secondary Outcome: Voice Quality Index 2: Acoustic Voice Quality Index (AVQI)
Description: A lower AVQI indicates a better voice quality. The index ranges from 0 to 10 for normal to severely dysphonic voices. An AVQI of 2.95 is the threshold separating normophonic from dysphonic persons.
Time Frame: baseline (before the intervention), 1 month (immediately after the intervention), 1 month follow-up, 3 months follow-up
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Straw Phonation in Air | Straw Phonation in 2 cm Water | Straw Phonation in 5 cm Water | /u/ Control Condition
Number analyzed (Participants) | 8 | 8 | 8 | 8
score on a scale
  baseline | 3.63 [3.07 to 4.20] | 3.69 [3.12 to 4.25] | 4.12 [3.56 to 4.69] | 3.70 [3.14 to 4.27]
  1 month | 3.86 [3.30 to 4.43] | 3.12 [2.56 to 3.69] | 3.73 [3.17 to 4.30] | 3.41 [2.84 to 3.97]
  1 month follow-up | 3.64 [3.08 to 4.21] | 3.22 [2.63 to 3.80] | 3.74 [3.17 to 4.30] | 3.57 [2.99 to 4.16]
  3 months follow-up | 3.84 [3.27 to 4.40] | 3.22 [2.64 to 3.81] | 3.86 [3.29 to 4.42] | 3.15 [2.53 to 3.76]

5. Secondary Outcome: Self-report 1: Voice Handicap Index (VHI)
Description: VHI: A lower index indicates less impact of the voice impairment on the quality of life. The VHI ranges from 0 to 120.
Time Frame: baseline (before the intervention), 1 month (immediately after the intervention), 1 month follow-up, 3 months follow-up
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Straw Phonation in Air | Straw Phonation in 2 cm Water | Straw Phonation in 5 cm Water | /u/ Control Condition
Number analyzed (Participants) | 8 | 8 | 8 | 8
score on a scale
  baseline | 9 [1 to 17] | 12 [4 to 20] | 19 [11 to 27] | 13 [5 to 20]
  1 month | 7 [0 to 15] | 12 [4 to 20] | 17 [9 to 24] | 13 [5 to 21]
  1 month follow-up | 9 [1 to 16] | 11 [3 to 19] | 18 [10 to 25] | 9 [1 to 17]
  3 months follow-up | 11 [3 to 19] | 16 [8 to 24] | 18 [10 to 25] | 11 [3 to 19]

6. Secondary Outcome: Self-report 2: Vocal Tract Discomfort Scale (VTDS)
Description: VTDS: A lower index indicates less discomfort in the vocal tract. The index ranges from 0 to 96.
Time Frame: baseline (before the intervention), 1 month (immediately after the intervention), 1 month follow-up, 3 months follow-up
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Straw Phonation in Air | Straw Phonation in 2 cm Water | Straw Phonation in 5 cm Water | /u/ Control Condition
Number analyzed (Participants) | 8 | 8 | 8 | 8
score on a scale
  baseline | 16 [7 to 25] | 21 [12 to 30] | 25 [16 to 34] | 16 [6 to 25]
  1 month | 13 [4 to 22] | 19 [10 to 28] | 21 [12 to 30] | 16 [7 to 25]
  1 month follow-up | 13 [3 to 22] | 16 [7 to 25] | 19 [10 to 28] | 21 [12 to 30]
  3 months follow-up | 13 [4 to 22] | 18 [9 to 27] | 20 [11 to 29] | 12 [2 to 21]

7. Secondary Outcome: Self-report 3: Vocal Fatigue Index (VFI)
Description: VFI: A lower index indicates less vocal fatigue. The index ranges from 0 to 76.
Time Frame: baseline (before the intervention), 1 month (immediately after the intervention), 1 month follow-up, 3 months follow-up
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Straw Phonation in Air | Straw Phonation in 2 cm Water | Straw Phonation in 5 cm Water | /u/ Control Condition
Number analyzed (Participants) | 8 | 8 | 8 | 8
score on a scale
  baseline | 14 [8 to 20] | 20 [14 to 26] | 19 [13 to 25] | 15 [9 to 21]
  1 month | 11 [5 to 17] | 14 [8 to 20] | 16 [10 to 22] | 15 [9 to 21]
  1 month follow-up | 11 [5 to 16] | 12 [6 to 18] | 17 [11 to 23] | 14 [8 to 20]
  3 months follow-up | 13 [7 to 19] | 17 [11 to 23] | 19 [13 to 25] | 15 [9 to 22]

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Straw Phonation in Air | Straw Phonation in 2 cm Water | Straw Phonation in 5 cm Water | /u/ Control Condition
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/13 | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13 | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 0/14 | 0/13 | 0/13 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-03): https://cdn.clinicaltrials.gov/large-docs/31/NCT06137131/Prot_SAP_000.pdf